CLINICAL TRIAL: NCT04281303
Title: Proof-of-concept Study of the Use of Endoscopic Gastroplasty in Patients With Obesity and Non-alcoholic Steatohepatitis Compensated Liver Cirrhosis (NASH)
Brief Title: Endoscopic Bariatric Therapy in NASH Cirrhosis
Acronym: ETHIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: ETHIC
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: NASH; Obesity; endoscopic vertical gastroplasty; cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic vertical gastroplasty: Proof-of-concept study that will prospectively include a number of patients undergoing endoscopic vertical gastroplasty + lifestyle modifications to evaluate the effect of this technique in an adult population with obesity and NASH cirrhosis
  Interventions: Procedure: Endoscopic vertical gastroplasty

INTERVENTIONS:
Procedure: Endoscopic vertical gastroplasty — endoscopic vertical gastroplasty + lifestyle modification

SUMMARY:
Non-alcoholic steatohepatitis (NASH) is a growing public health problem that affects more than 5% of the population and can lead to cirrhosis and hepatocellular carcinoma. These patients are at greater risk of cardiovascular and hepatic death, and higher rates of neoplasms, both gastrointestinal and extra-intestinal. The standard treatment is weight loss with diet and physical exercise, which has shown a histological and analytical improvement in patients who achieve a 5-10% reduction in body weight. However, less than 25% of subjects achieve this goal. Restrictive surgical treatments and gastric bypass have achieved, in obese patients, an improvement in metabolic syndrome, insulin resistance and liver histology, but in patients with liver cirrhosis the morbidity-mortality of this surgery is high. Currently, endoscopic techniques are being developed, which are less invasive and have fewer complications, and which also achieve gastric restriction with similar characteristics to those obtained by the surgical method. Among them is the tubulization or vertical gastroplasty with the OverStitch system (Apollo Endosurgery, Austin, TX, USA). However, this method has not been evaluated in patients with obesity and/or metabolic syndrome and NASH cirrhosis. For this reason, the main objective of the investigators study is to evaluate the safety and efficacy of endoscopic gastroplasty in improving metabolic factors and liver histology in patients with obesity with or without metabolic syndrome and NASH-compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects between the ages of 18 and 65 (inclusive) at the time of the first selection visit 2) They must provide a signed written informed consent and agree to comply with the study protocol.

  3) Subjects with a BMI greater than 30 kg/m2 whether or not associated with metabolic risk factors (MD, hypertension, dyslipemia).

  4) Confirmed diagnosis of non-alcoholic steatohepatitis with a degree of fibrosis 4 according to the NASH CRN staging system in a liver biopsy obtained in the 12 months prior to the endoscopic procedure or during the screening period.

  5) Absence of other causes of chronic liver disease (alcoholic, viral, autoimmune, cholestatic disease, Wilson's disease, α1AT deficit, hemochromatosis)

Exclusion Criteria:

1. Current or past history of any liver decompensation event (ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome, hepatopulmonary syndrome).
2. Child-Pugh Scale ≥ 7 points.
3. MELD scale > 12
4. Documented presence of varicose veins based on a previous endoscopy performed in the 6 months prior to the intervention.
5. Documented presence of collateral circulation based on an echoendoscopy and/or thoraco-abdominal CT with 3D reconstruction performed in the selection period.
6. Presence of a hepatic venous pressure gradient (HVPG) ≥ 10 mmHg in a hemodynamic study performed in the 4 months prior to surgery or in the selection period.
7. Known heart failure (Grade I-IV of the New York Heart Association classification).
8. History of bariatric surgery
9. Patients with a history of clinically significant cardiovascular events in the 6 months prior to the endoscopic procedure, such as an acute cardiovascular event, stroke, transient ischemic attack, or coronary heart disease (angina, myocardial infarction, revascularization procedures).
10. Weight loss of more than 5 % in the 6 months prior to the operation.
11. Recent or current history of significant consumption of alcoholic beverages (< 5 years) For men, significant consumption is usually defined as more than 30 g of pure alcohol per day. For women, it is normally defined as more than 20 g of pure alcohol per day.
12. Hepatocarcinoma. (13) Portal thrombosis.

14) Pregnancy. 15) Refusal to give informed consent. 16) Any medical condition that could reduce life expectancy to less than 2 years, including known cancers.

17) Indications of any other untreated, unstable or clinically significant immunological, endocrine, haematological, gastrointestinal, neurological, neoplastic or psychiatric disease.

18) Mental instability or incompetence such that the validity of the informed consent or the ability to comply with the study is uncertain.

19) Positive antibodies to human immunodeficiency virus. 20) Data on decompensated liver disease:

1. Aspartate aminotransferase (AST) and/or ALT > 10 x upper limit of normality (LSN)
2. Total bilirubin > 2 mg/dL
3. International Normalized Ratio (INR) > 1,4
4. Platelet count ≤ 100 000/mm3.
5. Albumin < 3.5 g/dL. 21) Serum creatinine levels > 135 μmol/l (> 1.53 mg/dl) in men and > 110 μmol/l (> 1.24 mg/dl) in women 22) Significant renal disease, including nephrotic syndrome, chronic renal disease (patients with markers of liver injury or estimated glomerular filtration rate [eGFR] of less than 60 ml/min/1.73 m2). If an abnormal value is obtained at the first screening visit, eGFR measurement may be repeated before randomisation within the following time frame: minimum 4 weeks after the initial test and maximum 2 weeks before the intended randomisation. Repeated abnormal eGFR (less than 60 ml/min/1,73 m2 ) leads to exclusion from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given the lack of previous studies on the efficacy of this technique in this type of patient, this proof-of-concept study will include a relatively small number of patients in order to obtain safety data and preliminary estimates of efficacy.
  Patients must present with obesity (BMI ≥ 30) associated or not with a metabolic syndrome according to NCEP ATP III criteria, which is already an indication for endoscopic treatment, and the diagnosis of cirrhosis by NASH according to histology (See inclusion criteria), which is a relative contraindication for the performance of bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Number of adverse events resulting from the procedure during the study
To evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Number of events related to liver disease: ascites, bleeding secondary to PTH, encephalopathy, SBP, or renal failure
To evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Number of cardiovascular events during follow-up: Ischemic heart disease, stroke, peripheral arterial disease, heart failure, cardiomyopathy.
Number of the patients to evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Death from all causes
Number of the patients to evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Liver transplant
Number of the patients to evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Model for end-stage liver disease (MELD) ≥ 15.
To evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Worsening of the Child-Pugh score by at least 2 points
Number of the patients to evaluate the safety of endoscopic vertical gastroplasty + lifestyle modification | 96 weeks
  Appearance of hepatocellular carcinoma (HCC)
To evaluate the efficacy of endoscopic vertical gastroplasty + lifestyle modification in the histological improvement of fibrosis | 96 weeks
  using the percentage of subjects with improvement in at least 1 stage in fibrosis without worsening of NASH

SECONDARY OUTCOMES:
Evaluate the following histological changes of treatment according to NASH-CRN criteria | after 96 weeks
  Changes in fibrosis including: improvement, not worsening, and progression
Evaluate the following histological changes of treatment according to NASH-CRN criteria | after 96 weeks
  Resolution of NASH defined as the presence or not of steatosis, without ballooning and with no or minimal inflammation.
Reduction the following histological changes of treatment according to NASH-CRN criteria | after 96 weeks
  Improvement of at least 1 point in the different components of the NASH-CRN score (steatosis, liver ballooning, and lobular inflammation)
Evaluate the following histological changes of treatment according to NASH-CRN criteria | after 96 weeks
  Improvement of fibrosis in at least 1 stage along with NASH improvement, defined as at least 1 stage improvement in fibrosis and at least 2 points less in NAFLD activity score (NAS) with at least 1 point improvement in ballooning and lobular swelling.
Evaluate the following histological changes of treatment according to NASH-CRN criteria | after 96 weeks
  NAS score changes.